CLINICAL TRIAL: NCT00578201
Title: Phase II Trial of FOLFOX in Combination With Cetuximab and Concomitant Radiotherapy in the Treatment of Esophageal Cancer Stage III
Brief Title: FOLFOX-Cetuximab-radiotherapy for the Treatment of Esophageal Cancer
Acronym: FOLFOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Isabelle BRINDEL, Departement clinical research of the developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P060503
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2007-05

CONDITIONS: Esophageal Cancer Stage III
Keywords: Esophageal neoplasms; Cetuximab; Oxaliplatin; Fluorouracil; radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): radiochemotherapy,combination Cetuximab-FOLFOX
  Interventions: Drug: radiochemotherapy,combination Cetuximab-FOLFOX

INTERVENTIONS:
Drug: radiochemotherapy,combination Cetuximab-FOLFOX — objective response rate at 12 weeks with radiochemotherapy then combination Cetuximab-FOLFOX
  Other Names: objective response rate,combination Cetuximab-FOLFOX

SUMMARY:
This phase II trial is studying the effects of oxaliplatin, leucovorin and fluorouracil-when given together with Cetuximab and radiation therapy and radiation therapy to see how they work in treating patients with stage III esophageal cancer.

DETAILED DESCRIPTION:
Cetuximab is a monoclonal antibody which can block the ability of tumor cells to grow and spread Cetuximab may also make tumor cells more sensitive to radiation therapy. Drug used in chemotherapy such as oxaliplatin leucovorin and Fluorouracil work in different way to stop the growth of tumor cells either by killing the cells or by stopping them form dividing. Radiation therapy uses high energy X rays to kill tumor cells. Giving cetuximab could improve the efficacy of chemotherapy and radiation therapy and may make the tumor smaller This phase II trial is studying the effects of oxaliplatin, leucovorin and fluorouracil-when given together with Cetuximab and radiation therapy and radiation therapy to see how they work in treating patients with stage III esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the esophagus stage III (according to UICC classification)
* Measurable disease according to the RECIST criteria
* WHO performance status of 0 or 1
* Age 18-80 years old
* Reference imaging within the 2 weeks prior to the treatment
* Hematological and biochemical assessment within the 2 weeks prior to the treatment
* Neutrophils >1.5 10 9/L, platelets >150.10 9/L, Haemoglobin ≥10g/dL, Bilirubin ≤ 1.25 ULN, Aspartate Aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 ULN Woman of childbearing potential must use effective contraception methods Written informed consent obtained No prior chemotherapy or radiation therapy for esophageal cancer

Exclusion Criteria:

* Stage I, II or IV (according to UICC classification)
* Esophageal carcinoma with small cells or endocrine cells or esophageal stromal tumor
* visceral metastasis
* orotracheal fistula weight loss >15% within the previous 6 months Pregnancy or breast feeding Contra indication to the study treatment History of coronary heart disease uncontrolled, or myocardial necrosis within the previous 6 months
* Peripheral Neuropathy NCI >1
* Liver Failure
* Prior thoracic radiation therapy
* history of cancer within the previous 5 years (except removed skin carcinoma, removed local melanoma located, and carcinoma cervix of uterus Esophageal Endoprosthesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) at 12 weeks with radiochemotherapy (first evaluation), and if applicable, within 2 to 4 weeks following the end of additional treatment with the combination Cetuximab-FOLFOX (second evaluation) | at 12 weeks and within 2 to 4 weeks following the end of additionnal treatment

SECONDARY OUTCOMES:
Progression free survival Quality of life Dysphagia score Overall survival toxicity of this regimen | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Gérard LLEDO, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Clinique Saint Jean, Lyon, France